CLINICAL TRIAL: NCT04769908
Title: Systemic Chemotherapy With Oxaliplatin and 5-fluorouracil, Lenvatinib Plus Sintilimab for With Distant Metastasis: a Single Arm Prospective Study
Brief Title: Systemic Chemotherapy, Lenvatinib Plus Sintilimab for ICC With Distant Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-077C
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: ICC
Keywords: ICC; Lenvatinib; Sintilimab; Systemic Chemotheray
MeSH Terms: interventions — Neoadjuvant Therapy; lenvatinib; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systemic Chemotherapy, Lenvatinib Plus Sintilimab (Experimental)
  Interventions: Drug: Systemic Chemotherapy; Drug: Lenvatinib; Drug: Sintilimab

INTERVENTIONS:
Drug: Systemic Chemotherapy — Systemic Chemotherapy (Oxaliplatin#5-fluorouracil and leucovorin)
Drug: Lenvatinib — Lenvatinib, 8mg or 12mg, po, QD
Drug: Sintilimab — Sintilimab, IV, 200mg, q3w

SUMMARY:
This study were designed to verify the better method of survival for ICC with distant metastasis. Since the traditional method for ICC with distant metastasis. was GEMOX(first-line treatment from NCCN guideline), our previous study found similar results from FOLFOX (second-line treatment from NCCN guideline) compared with GEMOX.

Our current study were conducted for further investigation to verify the better method for with distant metastasis.

DETAILED DESCRIPTION:
ICC (Intrahepatic CholangioCarcinoma) patients with metastasis has a short survival time and poor prognosis after diagnosis. Treatment methods was few and far from satisfaction. The treatment recommended from NCCN guideline was GEMOX (Systemic Chemotheray) and clinical trials. Our previous study has demonstrate FOLFOX (Systemic Chemotheray based on Oxaliplatin#5- fluorouracil) has a similar survival and tumor response compared with GEMOX. Further study was needed to intensive confirmation of the result. We designed this study to demonstrate the hypothesis. Metastasis ICCs were recruited and screened by our criteria. All patients were treated with FOLFOX (Systemic Chemotheray based on Oxaliplatin#5-fluorouracil ), lenvatinib (one of tyrosine kinase inhibitors) plus sintilimab (one of PD-1 antibody).

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of Intrahepatic CholangioCarcinoma (ICC)
* With distant metastasis
* Patients must have at least one tumor lesion that can be accurately measured according to mRECIST criteria.
* With no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment
* The following laboratory parameters:

Platelet count ≥ 60,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/ L Serum albumin ≥ 32 g/L ASL and AST ≤ 6 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-23 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate per RECIST | 6 months
  complete response and partial response per RECIST

SECONDARY OUTCOMES:
Overall survival | 6 months
Progression-free survival | 6 months
Number of adverse events | 30 days
  Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China